CLINICAL TRIAL: NCT04006964
Title: Diagnostic Accuracy Of Forced Oscillation Technique To Detect Lung Function Anomalies
Status: Completed | Type: Observational
Sponsor: Restech Srl (Industry)
Collaborators: MGC Diagnostics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2/17
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Identification Group: Subjects >= 3 years old will measure as a minimum FOT and spirometry. Final diagnosis will be made by the physician as per current guidelines.
  Interventions: Device: Resmon PRO FULL v2
- Validation Group: Subjects >= 3 years old will measure as a minimum FOT and spirometry. Final diagnosis will be made by the physician as per current guidelines.
  Interventions: Device: Resmon PRO FULL v2

INTERVENTIONS:
Device: Resmon PRO FULL v2 — Measurement of lung impedance by the Forced Oscillation Technique

SUMMARY:
The diagnosis of a lung function anomaly requires the evaluation of pulmonary function by spirometry. However, some patients (e.g. children, elderly, or diseased individuals) may have difficulty performing the related forced maximal respiratory maneuver correctly. Forced Oscillation Technique (FOT) measures lung impedance during tidal breathing, requiring minimal patient cooperation. The purpose of this study is to establish the diagnostic accuracy of FOT parameters alone or in combination with lung volumes in detecting lung function anomalies as compared with spirometry and with the diagnosis made by the physician.

DETAILED DESCRIPTION:
Purpose and Rationale The diagnosis of a lung function anomaly requires the evaluation of pulmonary function by spirometry. However, some patients (e.g. children, elderly, or diseased individuals) may have difficulty performing the related forced maximal respiratory maneuver correctly. FOT measures lung impedance during tidal breathing, requiring minimal patient cooperation. The within-breath calculation of impedance allows separating the contribution of inspiration and expiration to the measured parameters. The purpose of this study is to establish the diagnostic accuracy of FOT parameters alone or in combination with lung volumes in detecting lung function anomalies as compared with spirometry and with the diagnosis made by the physician.

Objectives Primary: To compare the diagnostic accuracy of FOT with spirometry to detect a lung function anomaly (i.e. an obstructive and/or restrictive respiratory disease).

Secondary: To compare the diagnostic accuracy of FOT with the final diagnosis made by the physician (i.e. the diagnosis based on current guidelines) to detect a lung function anomaly (i.e. an obstructive and/or restrictive respiratory disease).

Study Design This will be a multi-center prospective study of consecutive subjects attending the pulmonary function test laboratory for pulmonary function tests (PFT) or randomly taken from the clinical site's records among those with symptoms with two separate study phases, an Identification Phase and a Validation Phase. Subjects will undergo the same study procedures in both phases. After signing the Informed Consent, a medical history will be obtained, a physical examination performed, and PFT (FOT, spirometry and, if required by the physician to reach a final diagnosis, additional lung function measurements) will be performed.

Identification Phase: Subject data will be used to identify two separate rules based on abnormal lung volumes and impedance (FOT) parameters that will maximize the accuracy in identifying a lung function anomaly. For the primary objective, the reference test for the determination of such lung anomaly will be spirometry. For the secondary objective, the reference test for the determination of the presence of a lung function anomaly will be the final diagnosis made by the physician.

Validation Phase: A separate and independent dataset of subjects will be used to test the accuracy of the rules identified from analysis of the Identification Phase in detecting a lung function anomaly.

Study Duration Subject participation will be completed in 1 day. Study duration is expected to be 7 months

ELIGIBILITY:
Inclusion Criteria:

* All subjects ≥3 years old attending the pulmonary function laboratory with an order for PFT or
* Subjects ≥3 years old randomly chosen from a database of subjects having respiratory symptoms at the time of inclusion into the database.

Exclusion Criteria:

- Subjects unable to provide written Informed Consent (or not provided by the participant's parent/guardian) and Assent Form (where applicable).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The following age groups will be considered:
  * Preschool children (3-5 years old)
  * School-age children (6-11 years old)
  * Adolescents (12-17 years old)
  * Adults (>= 18 years old)
Sampling Method: Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-06-26 (Actual)

PRIMARY OUTCOMES:
Decision rule that maximises sensitivity and specificity as compared with spirometry | 1 day
  This will be a rule to detect lung anomalies as compared with spirometry that will be identified and validated in two separate populations

SECONDARY OUTCOMES:
Decision rule that maximises sensitivity and specificity as compared with physician's diagnosis | 1 day
  This will be a rule to detect lung anomalies as compared with physician's final diagnosis that will be identified and validated in two separate populations

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Inchingolo, MD, Principal Investigator — Catholic University of the Sacred Heart; Stefania La Grutta, MD, Principal Investigator — Istituto di Biomedicina e Immunologia Molecolare "A. Monroy"; Enrico Lombardi, MD, Principal Investigator — Meyer Children's Hospital IRCCS; David Kaminsky, MD, Principal Investigator — University of Vermont Medical Center Inc; Janos Porszasz, MD, Principal Investigator — Biomedical Research Institute at Harbor- UCLA Medical Center
Locations (6):
- United States (2):
  - Biomedical Research Institute at Harbor- UCLA Medical Center, Los Angeles, California
  - University of Vermont Medical Center Inc.,, Burlington, Vermont
- Italy (4):
  - Azienda Ospedaliero, Universitaria Meyer, Florence, FI
  - Catholic University of the Sacred Heart, Rome, Lazio
  - ASST Papa Giovanni XXIII, Bergamo
  - Istituto di Biomedicina e Immunologia Molecolare "A. Monroy", Palermo

REFERENCES:
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Aurora P, Stocks J, Oliver C, Saunders C, Castle R, Chaziparasidis G, Bush A; London Cystic Fibrosis Collaboration. Quality control for spirometry in preschool children with and without lung disease. Am J Respir Crit Care Med. 2004 May 15;169(10):1152-9. doi: 10.1164/rccm.200310-1453OC. Epub 2004 Mar 17. PMID 15028561
- [Background] Woodruff PG, Barr RG, Bleecker E, Christenson SA, Couper D, Curtis JL, Gouskova NA, Hansel NN, Hoffman EA, Kanner RE, Kleerup E, Lazarus SC, Martinez FJ, Paine R 3rd, Rennard S, Tashkin DP, Han MK; SPIROMICS Research Group. Clinical Significance of Symptoms in Smokers with Preserved Pulmonary Function. N Engl J Med. 2016 May 12;374(19):1811-21. doi: 10.1056/NEJMoa1505971. PMID 27168432
- [Background] van Noord JA, Wellens W, Clarysse I, Cauberghs M, Van de Woestijne KP, Demedts M. Total respiratory resistance and reactance in patients with upper airway obstruction. Chest. 1987 Sep;92(3):475-80. doi: 10.1378/chest.92.3.475. PMID 3622024
- [Background] Zerah F, Lorino AM, Lorino H, Harf A, Macquin-Mavier I. Forced oscillation technique vs spirometry to assess bronchodilatation in patients with asthma and COPD. Chest. 1995 Jul;108(1):41-7. doi: 10.1378/chest.108.1.41. PMID 7606989
- [Background] Faria AC, Costa AA, Lopes AJ, Jansen JM, Melo PL. Forced oscillation technique in the detection of smoking-induced respiratory alterations: diagnostic accuracy and comparison with spirometry. Clinics (Sao Paulo). 2010;65(12):1295-304. doi: 10.1590/s1807-59322010001200012. PMID 21340218
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Background] Dellaca RL, Aliverti A, Lo Mauro A, Lutchen KR, Pedotti A, Suki B. Correlated variability in the breathing pattern and end-expiratory lung volumes in conscious humans. PLoS One. 2015 Mar 24;10(3):e0116317. doi: 10.1371/journal.pone.0116317. eCollection 2015. PMID 25803710
- [Background] Peslin R, Ying Y, Gallina C, Duvivier C. Within-breath variations of forced oscillation resistance in healthy subjects. Eur Respir J. 1992 Jan;5(1):86-92. PMID 1577156
- [Background] Dellaca RL, Pompilio PP, Walker PP, Duffy N, Pedotti A, Calverley PM. Effect of bronchodilation on expiratory flow limitation and resting lung mechanics in COPD. Eur Respir J. 2009 Jun;33(6):1329-37. doi: 10.1183/09031936.00139608. Epub 2009 Jan 22. PMID 19164347
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Beydon N, Davis SD, Lombardi E, Allen JL, Arets HG, Aurora P, Bisgaard H, Davis GM, Ducharme FM, Eigen H, Gappa M, Gaultier C, Gustafsson PM, Hall GL, Hantos Z, Healy MJ, Jones MH, Klug B, Lodrup Carlsen KC, McKenzie SA, Marchal F, Mayer OH, Merkus PJ, Morris MG, Oostveen E, Pillow JJ, Seddon PC, Silverman M, Sly PD, Stocks J, Tepper RS, Vilozni D, Wilson NM; American Thoracic Society/European Respiratory Society Working Group on Infant and Young Children Pulmonary Function Testing. An official American Thoracic Society/European Respiratory Society statement: pulmonary function testing in preschool children. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1304-45. doi: 10.1164/rccm.200605-642ST. No abstract available. PMID 17545458
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736
- [Background] Brazzale DJ, Hall GL, Pretto JJ. Effects of adopting the new global lung function initiative 2012 reference equations on the interpretation of spirometry. Respiration. 2013;86(3):183-9. doi: 10.1159/000352046. Epub 2013 Aug 14. PMID 23949369
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: An Updated List of Essential Items for Reporting Diagnostic Accuracy Studies. Clin Chem. 2015 Dec;61(12):1446-52. doi: 10.1373/clinchem.2015.246280. Epub 2015 Oct 28. PMID 26510957
- [Background] Senn S. Review of Fleiss, statistical methods for rates and proportions. Res Synth Methods. 2011 Sep;2(3):221-2. doi: 10.1002/jrsm.50. Epub 2011 Dec 14. No abstract available. PMID 26061787
- See also: Global Initiative for Asthma. Global strategy for asthma management and prevention, 2017. — http://ginasthma.org